CLINICAL TRIAL: NCT01460836
Title: Indirect Comparison of Tobramycin Solution for Inhalation Versus Aztreonam Lysine for Inhalation in the Treatment of Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: HEORUS0017
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Inhalation

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Tobramycin Solution
  Interventions: Drug: Tobramycin solution for inhalation
- Aztreonam lysine
  Interventions: Drug: Aztreonam lysine for inhalation

INTERVENTIONS:
Drug: Tobramycin solution for inhalation
  Groups: Tobramycin Solution
Drug: Aztreonam lysine for inhalation
  Groups: Aztreonam lysine

SUMMARY:
Matching-adjusted indirect comparison of tobramycin solution (TIS) versus aztreonam lysine (AZLI) using TIS patient level clinical trial data and AZLI aggregated clinical trial data from published literature.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 6 years of age with a documented Cystic fibrosis (CF) diagnosis,
* moderate-to severe lung disease,
* the ability to perform reproducible pulmonary function tests,
* Pseudomonas aeruginosa (PA) airway infection.

Exclusion Criteria:

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cystic fibrosis
Sampling Method: Non-Probability Sample
Dates: Start 2010-04; Primary Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Mean relative change in Forced Expiratory Volume in 1 second (FEV1) from baseline | Baseline, Weeks 2, 4 and 6

SECONDARY OUTCOMES:
Mean change in the density of Pseudomonas aeruginosa (PA) from baseline | Baseline, Weeks 2, 4 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals